CLINICAL TRIAL: NCT00273520
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Telithromycin 800 mg (Once Daily for 10 Days) as a Supplement to the Standard of Care for Patients With Acute Exacerbations of Asthma
Brief Title: TELICAST : Telithromycin in Acute Exacerbations of Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR3647A_3503
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — telithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Telithromycin

SUMMARY:
Primary Objective:

* The primary objective is to evaluate the clinical efficacy of telithromycin versus placebo as a supplement to the usual standard of care during an acute exacerbation of asthma. Efficacy will be assessed by:

  * Changes in the diary card summary symptom score assessed daily for 6 weeks, and
  * Changes in the domiciliary morning Peak Expiratory Flow Rate (PEFR) following oral telithromycin treatment

Secondary Objectives:

The secondary objectives of the study are:

* To evaluate the microbial activity of telithromycin during an exacerbation of asthma by:

  * Assessment of the patient's clinical improvement relative to initial C. pneumoniae or M. pneumoniae status, and
  * Analysis of the quantitative changes from baseline in C. pneumonia or M. pneumoniae by culture and quantitative Polymerase Chain Reaction (PCR).
* To evaluate the safety of 10 days of oral telithromycin as a supplement to the standard of care for patients with acute exacerbations of asthma
* To assess additional efficacy endpoints and health outcome evaluations following 10 days of treatment with either oral telithromycin or placebo, with either treatment used as a supplement to the standard of care for patients with acute exacerbations of asthma:

  * Changes and daily variability in the PEFR during the 6 weeks of study treatment,
  * Health status at follow-up (6 weeks)
  * Pulmonary function tests:

    * Forced Expiratory Volume in 1 second (FEV1)
    * Forced Vital Capacity (FVC)
    * Forced Expiratory Flow Rate (FEF25-75%)
  * Need for additional medications (e.g., inhaled corticosteroids, oral corticosteroids, bronchodilator use),
  * Time to next acute exacerbation of asthma.

ELIGIBILITY:
Inclusion criteria

Patients meeting all of the following criteria will be considered for enrollment in the study:

* A documented history of asthma for >6 months
* Presenting within 24 hours of initial medical care in an urgent care clinic, emergency room, or in-patient hospital setting. To qualify for enrollment they must present with the following signs and symptoms of an acute deterioration in asthma control: (reduced PEFR, increased wheeze, and dyspnea, with or without cough).
* A PEFR less than 80% of predicted normal
* Females who meet the following conditions:

  * postmenopausal for at least 1 year, or
  * surgically incapable of bearing children, or
  * of childbearing potential, and all of the following conditions are met:

    * had a normal menstrual flow within 1 month before study entry and
    * has a negative pregnancy test (serum b-subunit human chorionic gonadotropin [hCG]) immediately before study entry and
    * must agree to abstinence or use of an accepted method of contraception

Exclusion criteria

Patients presenting with any of the following will not be included in the study:

* Requiring immediate placement in an Intensive Care Unit
* Obvious known allergic precipitant for this episode of acute severe asthma (e.g., acute exposure to animal dander)
* Pneumonia
* Known long QT syndrome or familial history of long QT syndrome (if no previous electrocardiogram [ECG] has invalidated this risk factor), or personal history of coronary disease, ventricular arrhythmia, bradycardia <50 beats/min, or known uncorrected hypokalemia or magnesemia
* Known impaired hepatic or renal function
* Known diagnosis of myasthenia gravis
* Active or quiescent tuberculosis infections of the respiratory tract
* Acute exacerbation of chronic bronchitis, chronic obstructive pulmonary disease, cystic fibrosis, or emphysema
* A history of smoking of 10 pack-years or more
* Women who are breast feeding or are pregnant, as demonstrated by serum or urine pregnancy tests
* Suspected or known hypersensitivity to, or suspected serious adverse reaction to the macrolide class of antibiotics
* A concomitant condition (including clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease) that would make implementation of the protocol or interpretation of the study results difficult
* A recent (within the previous 3 months) history of alcohol or recreational drug misuse.
* Immunocompromised patients, including but not limited to:

  * patients with known human immunodeficiency virus (HIV) infection and have either had or have an AIDS defining condition (e.g., Kaposi's sarcoma, Pneumocystis carinii pneumonia) or a CD4 + T lymphocyte count of <200/mL
  * patients with neutropenia (<1500 neutrophils/mm3)
  * patients with metastatic or hematological malignancy
  * splenectomized patients or patients with known hyposplenia or asplenia
* Planned surgical treatment at any time during the course of the study that would be incompatible with the objectives of this study
* Other disease conditions or infections that could interfere with the evaluation of study treatment efficacy or safety
* Oral steroid-dependent asthma
* Antibiotic use within 30 days prior to enrollment
* Treated within 2 weeks prior to inclusion with CYP3A4 inducers such as rifampicin, phenytoin, carbamazepine, and St. John's Wart
* Currently receiving medication known to prolong QT interval such as cisapride, pimozide, astemizole and terfenadine, or potent CYP3A4 inhibitors such as antiproteases or ketoconazole.
* Patients in whom an antibiotic is clearly indicated.
* Have received treatment with any other investigational drug within 1 month prior to study entry, or have such treatment planned for the study period during treatment and follow-up phase

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2003-01; Primary Completion 2004-04 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Patient's daily diary summary symptom scores/Morning diary PEFR | During the Study Conduct

SECONDARY OUTCOMES:
In-clinic pulmonary function tests: Forced expiratory volume in 1 second (FEV1), Percent predicted FEV1, Forced vital capacity (FVC), Forced expiratory flow rate at 25% to 75% of FVC (FEF25-75), PEFR, and percent predicted PEFR | During the study conduct
Evening diary PEFR, and diary PEFR variability | During the study conduct
Time to symptom resolution from study entry acute exacerbation of asthma | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, Study Director — Sanofi

REFERENCES:
- [Result] Johnston SL, Blasi F, Black PN, Martin RJ, Farrell DJ, Nieman RB; TELICAST Investigators. The effect of telithromycin in acute exacerbations of asthma. N Engl J Med. 2006 Apr 13;354(15):1589-600. doi: 10.1056/NEJMoa044080. PMID 16611950